CLINICAL TRIAL: NCT02812004
Title: New Horizons in the Treatment of Vitreous Floaters: Efficacy and Safety of Vitreolysis With the Ultra Q Reflex YAG Laser (Ellex)
Brief Title: New Horizons in the Treatment of Vitreous Floaters
Acronym: Ellex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AO Form 01-05/1.0 - Ellex
Record Dates: First submitted 2016-06-17; First posted 2016-06-23 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Other Vitreous Opacities, Bilateral
Keywords: Vitreous Floaters; Mouches Voulantes
MeSH Terms: conditions — vitreous floaters

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Eye (Experimental): Ultra Q Reflex YAG laser (Ellex)
  Interventions: Device: Ultra Q Reflex YAG laser (Ellex)
- Contralateral Eye (Sham Comparator): Short light impulse is simulated
  Interventions: Device: Ultra Q Reflex YAG laser (Ellex)

INTERVENTIONS:
Device: Ultra Q Reflex YAG laser (Ellex) — Group 1 receives up to 2 sessions of vitreolysis performed with the Ultra Q Reflex YAG laser (Ellex). There is no cut off for total energy per treatment session.
  For the sham treatment in group 2, the physician quickly manipulates the light switch of the laser's slit lamp to create light flashes and simulate laser pulses.

SUMMARY:
The Ultra Q Reflex® (Ellex) constitutes the only Nd:YAG laser approved for the treatment of vitreous floaters. No randomized controlled clinical trial has been carried out to this day in order to investigate its superiority over sham treatment.

In the present study, 60 eyes will be randomized and blinded into 2 groups, one receiving up to two sessions of laser vitreolysis the other scheduled for two sessions of sham treatment. After a maximum of two (sham) treatment sessions (1 per month), patients' utility value score and BCVA will be re-assessed. A follow-up period of 12 months (with visits at month 1, 6 and 12 post-treatment) will ensue the "treatment phase" to register any late adverse events that may be associated with laser vitreolysis.

As vitrectomy constitutes a highly invasive procedure, which must therefore be restricted to severe cases only, laser vitreolysis may present a valuable treatment option for patients with moderate vitreous floaters that are not eligible for vitrectomy.

DETAILED DESCRIPTION:
A great number of patients seek out their ophthalmologists when troubled by vitreous floaters. The majority of these patients are reassured when the diagnosis is made and are content to get accustomed to these "mouches volantes". A considerable proportion, however, feels permanently irritated by vitreous floaters which may result in a significant decrease of patients' quality of life.

Until recently, pars plana vitrectomy constituted the only established therapeutic option. Though a standard surgical procedure, the potential adverse events associated with vitrectomy are not negligible and patients must allow for an extended period of visual rehabilitation. Therefore, treatment was restricted to severe cases and thus only a very small percentage of patients received any treatment at all.

Reports exist on Q-switched Nd:YAG laser surgery for vitreous opacities, membranes and vitreoretinal bands in 59 eyes. The results of early laser vitreolysis are sobering with an improve in visual acuity in only 18 eyes but considerable adverse events such as retinal holes with detachment (1 eye), minor retinal hemorrhages (4 eyes) and focal opacities of the crystalline lens (5 eyes).

According to another study, the Q-switched system allowed treatment of a wider variety of indications in the posterior pole and requires fewer sessions when compared to a mode-locked system. Due to the higher energy levels required by Q-switch system, however, complications occurred more frequently.

An additional study presented more favorable results; in all 15 cases the symptoms of vitreous floaters disappeared after treatment and no adverse events were reported during a follow-up period of at least 1 year. Nevertheless, the reported energy levels (5-7.1mJ and total energy 71-742mJ) were considerable.

Further results suggested that laser vitreolysis moderately improved symptoms in 38% of all patients, while 61,5% registered no improvement; no adverse events were reported. In contrast, vitrectomy resulted in full resolution of symptoms in 93,3% of eyes - with one patient suffering post-operative retinal detachment.

A recent study presented 3 cases of chronic open-angle glaucoma secondary to ND:YAG vitreolysis (3 eyes of 2 patients). The latency period between vitreolysis and onset of elevated IOP ranged from 1 week to 8 months; other potential factors promoting a rise in IOP, namely "inflammation, steroid use, or other identifiable causes" are reported as absent. In two eyes, SLT followed by glaucoma surgery (Trabectome) was required to stabilise IOP.

Whereas the treatment of floaters located in the anterior vitreous resulted in no obvious change, treatment in the mid-vitreous and posterior vitreous lead to an increase in protein, the refractive index and the viscosity of the vitreous humor.

It appears that the current literature remains inconclusive as to the efficacy and safety of Nd:YAG vitreolysis. In the review literature, floater vitrectomy - especially with small sutureless gauge instruments and a corevitrectomy - yields excellent success rates combined with a low risk profile. In contrast, the efficacy of vitreolysis ranges between 0 and 100%. The key factor to success in vitreolysis is the use of appropriately high energy levels and the application of a sufficient amount of shots. In his retrospective, observational study (including 168 eyes, treatment with the Ultra Q Relfex®) 92% of patients were satisfied with the result;

In the present study, vitreolysis is performed with the Ultra Q Reflex® laser - to this day the only laser officially approved for vitreolysis. It features an ultra-Gaussian beam mode, teamed with a fast-pulse rise time and a small-spot size. Due to the tightly controlled plasma with its higher power density fewer shots are required which results in a lower cumulative dose. Moreover, the co-axial alignment of the practitioner's vision, the target illumination, and the treatment beam grants better illumination of vitreous opacities and thus allows for more precise focusing. This patented design facilitates the vaporization of floaters and minimizes the risk of collateral damage to adjacent tissues.

ELIGIBILITY:
Inclusion Criteria:

* the subject's written consent to participate in the present study
* considerable impairment of quality of life (defined as utility value score ≤ 0.7) due to floater-related symptoms for at least 3 months prior to inclusion
* floaters must be located at a safe distance to both the retina and the intraocular lens - preferably in the middle third of the vitreous
* pseudophakic eyes
* age >18 years

Exclusion Criteria:

* phakic eyes
* any retinal pathology and/or other ocular condition (including but not limited to amblyopia, pathologies of the cornea, glaucoma/history of elevated intraocular pressure) that may prevent or reduce a potential increase in visual acuity and/or decrease of the utility value score and/or incur an increased likelihood of adverse events.
* any ocular or systemic condition that may result in an impaired feasibility of the study treatment and/or required examinations.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Utility Value Score | 1-6 months
  Subjective Assessment of Impairment due to floaters

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ring, Dr, Study Director — Department of Ophthalmology
Locations (1):
- AKh Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Little HL, Jack RL. Q-switched neodymium: YAG laser surgery of the vitreous. Graefes Arch Clin Exp Ophthalmol. 1986;224(3):240-6. doi: 10.1007/BF02143063. PMID 3754829
- [Background] Tassignon MJ, Kreissig I, Stempels N, Brihaye M. Indications for Q-switched and mode-locked Nd: YAG lasers in vitreoretinal pathology. Eur J Ophthalmol. 1991 Jul-Sep;1(3):123-30. doi: 10.1177/112067219100100304. PMID 1841668
- [Background] Delaney YM, Oyinloye A, Benjamin L. Nd:YAG vitreolysis and pars plana vitrectomy: surgical treatment for vitreous floaters. Eye (Lond). 2002 Jan;16(1):21-6. doi: 10.1038/sj.eye.6700026. PMID 11913884
- [Background] Cowan LA, Khine KT, Chopra V, Fazio DT, Francis BA. Refractory open-angle glaucoma after neodymium-yttrium-aluminum-garnet laser lysis of vitreous floaters. Am J Ophthalmol. 2015 Jan;159(1):138-43. doi: 10.1016/j.ajo.2014.10.006. Epub 2014 Oct 13. PMID 25308785
- [Background] Abdelkawi SA, Abdel-Salam AM, Ghoniem DF, Ghaly SK. Vitreous humor rheology after Nd:YAG laser photo disruption. Cell Biochem Biophys. 2014 Mar;68(2):267-74. doi: 10.1007/s12013-013-9706-5. PMID 23797611